CLINICAL TRIAL: NCT01402167
Title: Evaluating Transcutaneous Vertebroplasty and Kyphoplasty for Reducing Trauma-related Fractures: a Randomized Pilot Study Using Catscan Volumetry
Brief Title: Evaluating Vertebroplasty and Kyphoplasty for Reducing Trauma-related Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients refuse randomization.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOCAL/2011/PK-04
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Vertebral Body Compression Fractures
MeSH Terms: interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kyphoplasty (Experimental): Patients randomized to this arm will be treated via balloon kyphoplasty.
  Interventions: Procedure: Kyphoplasty
- Vertebroplasty (Active Comparator): Patients randomized to this arm will be treated via vertebroplasty.
  Interventions: Procedure: Vertebroplasty

INTERVENTIONS:
Procedure: Kyphoplasty — Patients will be treated via a balloon kyphoplasty surgical procedure
  Arms: Kyphoplasty
Procedure: Vertebroplasty — Patients will be treated via a transcutaneous vertebroplasty procedure.
  Arms: Vertebroplasty

SUMMARY:
The primary objective of this study is to compare the volume of injected ciment (polymethyl methacrylate) between a group of patients treated with vertebroplasty and a group of patients treated via kyphoplasty. Secondary evaluation will compare the restoration of vertebral height, volume and cyphotic angle between the two techniques, as well as extravation of ciment and functional and quality of life aspects related to these techniques.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow-up
* Fracture type according to Magerl Classification (1994) must be one of the following: A1, A2.1, A3.1, A3.2
* Cyphose of >10°
* Spinal pain
* Vertebral fracture < 3 weeks old located between D5 and L5
* If fragments in the canal, they must protrude less than 40%
* Absence of other lesions, including cancer

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient cannot read French
* Patient is pregnant or breast feeding
* Patient has a fracture on an adjacent vertebra
* Patient has a contra-indication for a treatment used in this study
* ASA class IV or V
* Patient has a neurological deficit
* Previous spinal surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The volume (cm^3) of injected ciment | Baseline (Day 0)
  The volume of injected ciment is measured by catscan extrapolated data.

SECONDARY OUTCOMES:
Recovery of vertebral volume (%) | Day 1 to Day 7
  Recovery of vertebral volume relative to theoretical volume based on neighboring vertebra.
Change from baseline of the cyphotic angle (°) | Days 1 to 7
  The number of degrees of change in the cyphotic angle of the corrected vertebra relative to baseline measurement (°)
Change from baseline of the cyphotic angle (°) | 1 month
  The number of degrees of change in the cyphotic angle of the corrected vertebra relative to baseline measurement (°)
Change from baseline of the cyphotic angle (°) | 3 months
  The number of degrees of change in the cyphotic angle of the corrected vertebra relative to baseline measurement (°)
Change from baseline in vertebral height (mm) | Days 1 to 7
  Change in vertebra height (mm) before and after surgery
Change from baseline in vertebral height (mm) | 1 month
  Change in vertebra height (mm) before and after surgery
Change from baseline in vertebral height (mm) | 3 months
  Change in vertebra height (mm) before and after surgery
Volume of ciment leakage (cm^3) | Day 1
  The volume of ciment leakage will be determined according to catscan data.
Change in Visual Analog Scale (0 to 10) for pain before and after surgery | Day 0 (post-op)
  Brute change in Visual Analog Scale (0 to 10) for pain before and after surgery
Change in Visual Analog Scale (0 to 10) for pain before and after surgery | 1 month
  Brute change in Visual Analog Scale (0 to 10) for pain before and after surgery
Change in Visual Analog Scale (0 to 10) for pain before and after surgery | 3 months
  Brute change in Visual Analog Scale (0 to 10) for pain before and after surgery
% Change in Visual Analog Scale (0 to 10) for pain before and after surgery | Day 0 (post-op)
  The percentage change (%) in Visual Analog Scale (0 to 10) for pain before and after surgery
% Change in Visual Analog Scale (0 to 10) for pain before and after surgery | 1 month
  The percentage change (%) in Visual Analog Scale (0 to 10) for pain before and after surgery
% Change in Visual Analog Scale (0 to 10) for pain before and after surgery | 3 months
  The percentage change (%) in Visual Analog Scale (0 to 10) for pain before and after surgery
The change in the ODI score before and after surgery | 3 months
  The change in the Oswestry Disability Index before and after surgery
The % change in the ODI score before and after surgery | 3 months
  The percentage change (%) in the Oswestry Disability Index before and after surgery
Change in SF-36 quality of life score before and after surgery | 1 month
  Change in SF-36 quality of life score before and after surgery
Change in SF-36 quality of life score before and after surgery | 3 months
  Change in SF-36 quality of life score before and after surgery
The % change in SF-36 quality of life score before and after surgery | 1 month
  Percentage change (%) in SF-36 quality of life score before and after surgery
The % change in SF-36 quality of life score before and after surgery | 3 months
  Percentage change (%) in SF-36 quality of life score before and after surgery
Change in FABQ score before and after surgery | 1 month
  Change in the Fear-Avoidance Beliefs Questionnaire score before and after surgery
Change in FABQ score before and after surgery | 3 months
  Change in the Fear-Avoidance Beliefs Questionnaire score before and after surgery
% Change in FABQ score before and after surgery | 1 month
  Percentage change (%) in the Fear-Avoidance Beliefs Questionnaire score before and after surgery
% Change in FABQ score before and after surgery | 3 months
  Percentage change (%) in the Fear-Avoidance Beliefs Questionnaire score before and after surgery
Change in DPQ score before and after surgery | 1 month
  Change in the Dallas Pain Questionnaire score before and after surgery
Change in DPQ score before and after surgery | 3 months
  Change in the Dallas Pain Questionnaire score before and after surgery
% Change in DPQ score before and after surgery | 3 months
  Percentage change (%) in the Dallas Pain Questionnaire score before and after surgery
% Change in DPQ score before and after surgery | 1 month
  Percentage change (%) in the Dallas Pain Questionnaire score before and after surgery
Duration of surgery (minutes) | Day 0 (day of surgery)
  Length of operative time (minutes)
Presence / absence of per-operative complications | Day 0 (day of surgery)
  Presence / absence of per-operative complications
Presence / absence of post-operative complications | 1 month
  Presence / absence of post-operative complications
Presence / absence of post-operative complications | 3 months
  Presence / absence of post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Kouyoumdjian, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes